CLINICAL TRIAL: NCT05074784
Title: Effects of IOPI on Swallowing Function and Functional Status in Geriatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khoo Teck Puat Hospital (Other)
Collaborators: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Choo Wan Ling, Senior Speech Therapist, Khoo Teck Puat Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021/00223
Record Dates: First submitted 2021-09-18; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into control group or intervention group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Tongue depressor exercise protocol for tongue strengthening for control group. Using the tongue depressor, participants will be prompted to stick their tongue out as much as they can and to push hard against the tongue depressor for 10 seconds. They will be required to repeat this action 10 times, constituting one set. They will be asked to perform 3 sets, with 30 secs of rest between each set. Arrange for 5 sessions for a week; sessions can take place on consecutive days.
  Interventions: Device: Tongue Depressor Traditional Intervention
- Intervention Group (Experimental): IOPI exercise protocol for tongue strengthening for intervention group. Using the IOPI, participants will perform 24 sets of 5 repetition at anterior position, allowing for 30 secs rest in between sets. Arrange for 5 sessions for a week; sessions can take place on consecutive days.
  Interventions: Device: IOPI Therapy

INTERVENTIONS:
Device: IOPI Therapy — Obtain IOPI reading at start of session, record the best of 3 readings as baseline strength. Calculate exercise resistance for session at 60% of baseline strength. Using the IOPI, participants will perform 24 sets of 5 repetition at anterior position, allowing for 30 secs rest in between sets.
  Arms: Intervention Group
Device: Tongue Depressor Traditional Intervention — Using the tongue depressor, participants will be prompted to stick their tongue out as much as they can and to push hard against the tongue depressor for 10 seconds. They will be required to repeat this action 10 times, constituting one set. They will be asked to perform 3 sets, with 30 secs of rest between each set
  Arms: Control Group

SUMMARY:
This project is an exploratory study that aims to investigate the effects of IOPI therapy on the swallowing function and tongue strength of geriatric patients in a geriatric ward in an acute hospital. Its secondary aim is to investigate the correlation between IOPI readings and functional status. The result of this study could help to improve current practice of dysphagia intervention in the geriatric population. If results are significant, there will be research evidence to put forth a change to work processes for speech therapists. IOPI will be more widely used in the clinical context and will then result in better functional outcomes.

DETAILED DESCRIPTION:
In recent years, there have been increasing evidence that tongue strengthening exercises have the ability to improve tongue muscle strength and tongue muscle thickness in the geriatric population. These improvements have a direct impact on the oral phase of swallow, specifically resulting in better orolingual manipulation and propulsion, and increasing intra-oral pressure for better bolus clearance. Reduction in tongue strength and other swallowing parameters can lead to swallowing disorder known as dysphagia. In the healthy ageing population, weakness in swallowing muscles is termed presbyphagia. Geriatric patients have an even higher chance of transitioning from presbyphagia to dysphagia when they become acutely unwell. Studies have also shown that deterioration of the whole-body muscle strength is associated with poorer oral function. Additionally, other studies have also shown that a lower isometric tongue strength might represent diminished functional reserves, which may increase the risk of dysphagia once an insult to the body occurs. There is also evidence that people who have episodes of aspiration have significantly weaker tongue strength at both the anterior and posterior regions. Thus, frail geriatric adults who have weaker skeletal muscles are at a higher risk of developing dysphagia. The tongue is amendable to therapy but current practices in Singapore lack an objective measure. Conventional dysphagia oromotor exercises employ the use of a tongue depressor. This method lacks a quantifiable measure to track outcome and is quite subjective to individual therapists. There is also a lack of practice guideline on recommended resistive load and frequency of exercise in the geriatric population in the acute setting. Other than outcome measures and practice guidelines, there is also a lack of research investigating the correlation of tongue strength and functional status. A few studies have explored the effects of different resistive load used in tongue strengthening exercises, although it was recommended to use a resistive load between 60% to 80% for more positive and extrinsic feedback, and for target population with a lower frustration threshold. Studies also used a longer timeframe of 3-4 weeks of rehabilitation to attain significant effects from skeletal muscle exercise. This, however, is not realistic in the acute geriatric setting in Singapore where the mean length of stay is 10 days. Thus, this study is an exploratory study to investigate the efficacy of using IOPI in this population to improve swallowing function and tongue strength. This study also aims to investigate if a correlation exists between IOPI reading and functional status.

ELIGIBILITY:
Inclusion Criteria:

1. aged 78-99 years old
2. CFS rating of 4-7
3. able to sit out of bed
4. able to follow at least 2-step directions (even for patients with cognitive condition e.g. dementia )
5. diagnosed with dysphagia by the ward speech therapist and assessed to be suitable for therapy
6. have not been admitted for more than 2 days

Exclusion Criteria:

1. acute neurological conditions such as traumatic brain injury or stroke
2. history of head and neck cancer, surgery or radiotherapy to head and neck region and 3) patients on long term tube feeding

Ages: 78 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of increase in tongue strength | 5 intervention days
  The IOPI device will be used to measure tongue strength at the anterior position on the last day of intervention. This will be compared to the baseline tongue strength collected on the first day of intervention.
Improvement in score on Functional Oral Intake Scale (FOIS) | 5 intervention days
  The speech therapist will rate the participant's FOIS score at the start and end of intervention according to the type of diet that the participant is prescribed.

SECONDARY OUTCOMES:
Improvement in AusTOMs Swallowing Scale Rating | 5 intervention days
  The speech therapist will rate the participant on the AusTOMs swallowing scale at the beginning and end of intervention with accordance to the severity of dysphagia.
Improvement in Modified Barthel Index (MBI) Score | 5 intervention days
  The occupational therapist will provide a baseline and outcome rating on the MBI for each participant. This will contribute to the evaluation of the patient's functional status at the end of intervention.
Improvement in hand grip strength (HGS) | 5 intervention days
  The speech therapist administering the intervention will assess for hand grip strength at the beginning and end of intervention. This will contribute to the evaluation of the patient's functional status at the end of intervention.
Improvement in timed sit-to-stand duration | 5 intervention days
  The speech therapist administering the intervention will assess for timed sit-to-stand at the beginning and end of intervention. This will contribute to the evaluation of the patient's functional status at the end of intervention.
Improvement in the score of the SARC-F questionnaire | 5 intervention days
  The speech therapist administering the intervention will complete the questionnaire with the participant at the beginning and end of intervention. This will contribute to the evaluation of the patient's functional status at the end of intervention.
Improvement in overall functional status. | 5 intervention days
  The investigators of the study will compare the baseline and outcome measures for the AusTOMs swallowing scale rating, MBI, HGS, timed sit-to-stand and SARC-F scores to evaluate if participants show an improvement in their overall functional status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams V, Mathisen B, Baines S, Lazarus C, Callister R. Reliability of measurements of tongue and hand strength and endurance using the Iowa Oral Performance Instrument with elderly adults. Disabil Rehabil. 2015;37(5):389-95. doi: 10.3109/09638288.2014.921245. Epub 2014 May 22. PMID 24854105
- [Background] Aoki, Y., Kabuto, S., Ozeki, Y., Tanaka, T., amp; Ota, K. (2015). The effect of tongue pressure strengthening exercise for dysphagic patients. Japanese Journal of Comprehensive Rehabilitation Science, 6, 129-136.
- [Background] Butler SG, Stuart A, Leng X, Wilhelm E, Rees C, Williamson J, Kritchevsky SB. The relationship of aspiration status with tongue and handgrip strength in healthy older adults. J Gerontol A Biol Sci Med Sci. 2011 Apr;66(4):452-8. doi: 10.1093/gerona/glq234. Epub 2011 Feb 7. PMID 21300744
- [Background] Kim, S., Kim, M., Lee, S., Choi, B., amp; Heo, Y. (2019). The Effects of Orofacial Myofunctional Training on the Changes of Lip and Tongue Strength in Elderly People. Journal of Dental Hygiene Science, 19(4), 279-287. doi:https://doi.org/10.17135/jdhs.2019.19.4.279
- [Background] Namasivayam-MacDonald AM, Riquelme LF. Presbyphagia to Dysphagia: Multiple Perspectives and Strategies for Quality Care of Older Adults. Semin Speech Lang. 2019 Jun;40(3):227-242. doi: 10.1055/s-0039-1688837. Epub 2019 Jun 3. PMID 31158906
- [Background] Park JS, Lee SH, Jung SH, Choi JB, Jung YJ. Tongue strengthening exercise is effective in improving the oropharyngeal muscles associated with swallowing in community-dwelling older adults in South Korea: A randomized trial. Medicine (Baltimore). 2019 Oct;98(40):e17304. doi: 10.1097/MD.0000000000017304. PMID 31577721
- [Background] Sagawa K, Furuya H, Ohara Y, Yoshida M, Hirano H, Iijima K, Kikutani T. Tongue function is important for masticatory performance in the healthy elderly: a cross-sectional survey of community-dwelling elderly. J Prosthodont Res. 2019 Jan;63(1):31-34. doi: 10.1016/j.jpor.2018.03.006. Epub 2018 Sep 7. PMID 30197226
- [Background] Van den Steen L, Schellen C, Verstraelen K, Beeckman AS, Vanderwegen J, De Bodt M, Van Nuffelen G. Tongue-Strengthening Exercises in Healthy Older Adults: Specificity of Bulb Position and Detraining Effects. Dysphagia. 2018 Jun;33(3):337-344. doi: 10.1007/s00455-017-9858-3. Epub 2017 Oct 19. PMID 29052051
- [Background] Van den Steen L, Vanderwegen J, Guns C, Elen R, De Bodt M, Van Nuffelen G. Tongue-Strengthening Exercises in Healthy Older Adults: Does Exercise Load Matter? A Randomized Controlled Trial. Dysphagia. 2019 Jun;34(3):315-324. doi: 10.1007/s00455-018-9940-5. Epub 2018 Sep 12. PMID 30209561
- [Background] Van den Steen L, De Bodt M, Guns C, Elen R, Vanderwegen J, Van Nuffelen G. Tongue-Strengthening Exercises in Healthy Older Adults: Effect of Exercise Frequency - A Randomized Trial. Folia Phoniatr Logop. 2021;73(2):109-116. doi: 10.1159/000505153. Epub 2020 Feb 5. PMID 32023617
- [Background] Yoshimi K, Nakagawa K, Hara K, Yamaguchi K, Nakane A, Kubota K, Furuya J, Tohara H. Relationship between tongue pressure and back muscle strength in healthy elderly individuals. Aging Clin Exp Res. 2020 Dec;32(12):2549-2555. doi: 10.1007/s40520-020-01484-5. Epub 2020 Jan 31. PMID 32006384
- [Background] Zhang H, Guo F, Tang M, Dai H, Sheng J, Chen L, Liu S, Wang J, Shi Y, Ye C, Hou G, Wu X, Jin X, Chen K. Association between Skeletal Muscle Strength and Dysphagia among Chinese Community-Dwelling Elderly Adults. J Nutr Health Aging. 2020;24(6):642-649. doi: 10.1007/s12603-020-1379-3. PMID 32510118